CLINICAL TRIAL: NCT04991909
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics of HRS4800 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS4800-103
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: HRS4800 Tablet compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: HRS4800
- Treatment group B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS4800 — HRS4800
  Arms: Treatment group A
Drug: Placebo — Placebo
  Arms: Treatment group B

SUMMARY:
The study is being conducted to assess the safety and tolerability of HRS4800 after multiple oral administration with different dose regimens in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Males and females aged between 18 years and 55 years at screening, inclusive.
3. Meet the weight standard
4. Agree to take effective contraceptive methods
5. No clinically significant abnormalities in medical history, general physical examination, vital signs, laboratory tests

Exclusion Criteria:

1. Severe infections, injuries or surgeries or plan to undergo any surgeries.
2. ALT, AST, ALP or total bilirubin level abnormal
3. Estimated Glomerular Filtration Rate (eGFR, using CKD-EPI Creatinine Equation) is abnormal
4. Subject's supine systolic BP is >140 mmHg or <90 mmHg; diastolic BP >90 mmHg or <40 mmHg at screening/baseline visits or before dosing.
5. Subjects with cardiac and Cerebrovascular Disease
6. Positive nicotine test
7. History of regular alcohol consumption in the past 1 month exceeding an average weekly intake of 21 standard drinks
8. Positive drug screening tests
9. Positive infectious diseases screening tests
10. plan to use of any other medicine during the trial
11. Whole blood donation or loss of more than 200 mL of blood within 1 month
12. blood transfusion in the past 2 months
13. History of allergy to the study drug or any component of it.
14. Can't accept assigned meals during the trial
15. Treatment with an investigational drug within 30 days (or 5 half-lives, whichever is longer) of dosing.
16. poor tolerance or difficult for vein blood collection
17. Other conditions or laboratory abnormality that may increase the risk associated with study participation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of the Adverse Events that are related to the treatment from baseline to Day36 | from baseline to Day36
The severity of the Adverse Events that are related to the treatment from baseline to Day36 | from baseline to Day36

SECONDARY OUTCOMES:
Cmax, Peak Concentration; | Day1
AUC0-tau, Area under the curve during a dose interval; | Day1
Tmax; The time to reach peak concentration; | Day1
Css,max, Peak Concentration at steady state; | Day14
AUCss, 0-tau, Area under the curve during a dose interval at steady state; | Day14
AUC0-inf, Area under the curve from 0 to infinite; | Day14
Tmax, the time to reach peak concentration; | Day14
Ctrough trough concentration at steady state; | Day14
Rac, , accumulation factor; | Day14
t1/2, terminal half life; | Day14
CL/F, apparent clearance at steady state ; | Day14
Vss/F; apparent volume of distribution at steady state | Day14
SHR175593 concentration on Day1 and day 14 | Day1 and day 14
QTc on Day1 and Day 14 | Day1 and day 14

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China